CLINICAL TRIAL: NCT02925962
Title: A Randomized Trial to Evaluate an Electronic CKD Clinical Decision Support System (CDSS) in Clinical Care
Brief Title: Evaluation of an Electronic CKD Clinical Decision Support System (CDSS) in Clinical Care
Acronym: CDSSR18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CP2016R18
Record Dates: First submitted 2016-09-30; First posted 2016-10-06 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Hypertension; Renal Insufficiency, Chronic
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical Decision Support System (CDSS) (Experimental): PCPs get a notice the CKD Clinical Decision Support System (CDSS) is available.
  CDSS overview:
  * The study MDs order CKD triple marker tests
  * Patients will go to the lab as per usual clinical care
  * Lab results are returned to PCPs clinical results folder as per usual clinical workflow with information about CKD and link to KDIGO guidelines
  * Results will also be sent to the Study MD's for monitoring
  * At the patient's next visit, if the labs are completed, the full CDSS launches for the PCP
  * If the labs are not completed by the next visit, a Best Practice Alert (BPA) will launch for the PCP notifying them that the labs have been ordered, but the patient hasn't done them yet
  Interventions: Other: Clinical Decision Support System (CDSS)
- Clinic Decision Sup System + Pharmacist (Experimental): The Clinical Decision Support System + Pharmacist follow-up call extends beyond the CDSS alone.
  CDSS Plus overview:
  * At the visit in which the CDSS launches, the PCP will hand a study card with pharmacist information to their patient notifying them that a pharmacist will be calling to follow-up after the visit
  * The pharmacist will use MyChart and/or phone calls to schedule a follow-up call within two weeks of the visit
  * On the follow-up phone call, the pharmacist will discuss understanding of CKD, medication review and adherence assessment, home BP checks, and the importance of NSAID avoidance
  * A second follow-up call will only be scheduled if the patient is non-adherent with their medications and makes an active plan for adherence with the pharmacist, or if the patient requests an additional call from the pharmacist
  Interventions: Other: Clinic Decision Sup System + Pharmacist
- Usual Care (No Intervention): Patients continue to receive usual care by their provider.

INTERVENTIONS:
Other: Clinical Decision Support System (CDSS) — A targeted, automated CKD clinical decision support system (CDSS) designed to improve bloodpressure (BP) level, disease awareness, staging, processes of care, and knowledge among persons with documented reduced eGFRcreat (creatinine-based estimated glomerular filtration rate) in primary care setting.
  Arms: Clinical Decision Support System (CDSS)
Other: Clinic Decision Sup System + Pharmacist — Includes everything in the CDSS intervention but adds a follow-up call from a pharmacist, who is part of the clinical team. The rationale for this third arm is based on the evidence that clinical pharmacists have been shown to be more effective than physicians alone at achieving BP control in other settings.
  Other Names: CDSS Plus, Clinical Decision Support System + Pharmacist
  Arms: Clinic Decision Sup System + Pharmacist

SUMMARY:
The investigators propose a three-arm, pragmatic, cluster-randomized clinical trial based in primary care. Participating Primary Care Providers (PCPs) will be randomized to usual care or one of two intervention arms. The first intervention will evaluate the efficacy of an automated CDSS that utilizes the electronic health record (EHR) to facilitate triple marker test ordering, guideline implementation and BP management, compared with usual care, among patients with previous documentation of eGFRcreat <60 ml/min/1.73m2. The second intervention goes a step further, and will evaluate whether a CDSS plus a follow-up telephone call from a pharmacist (CDSS PLUS) can improve BP management and patient CKD and NSAID toxicity knowledge among the patients with CKD, compared with CDSS alone. The primary clinical outcome is BP level, with secondary outcomes related to processes of care and patient knowledge.

DETAILED DESCRIPTION:
Setting:

The investigators will conduct this study within the three General Internal Medicine (GIM) practices at UCSF. These include general internal medicine PCPs who practice primary care. This trial is specifically designed to work within the framework of the existing infrastructure of these practices.

Randomization:

The unit for randomization will be the PCP (MD and NPs with their own panel of patients); the investigators plan to include up to 105 PCPs.

Training and Pre-Trial Preparation:

Prior to the beginning of this trial, all eligible providers at the UCSF GIM practice will be informed of this trial by the PI via email, attached with consent information, at which time they will be sent a link to information about the Kidney Disease Improving Global Outcomes (KDIGO) guidelines, and they will have the opportunity to opt-out of the trial. PCP randomization will be performed by the study coordinator using an automated procedure. The PCPs randomized to the intervention arms (CDSS and CDSS PLUS) will have the option to view a brief training video designed by study PIs and IT experts on the automated CKD CDSS.

Blinding:

The analysts will remain blinded throughout the trial and data analyses.

Intervention Details (CKD CDSS):

The CKD CDSS has been developed by the study PIs and IT experts, and refined using physician feedback. While the tool will be automated as much as possible using the electronic medical record, provider decision making will be required at all diagnostic or treatment steps in the CDSS.

The study MD will order all of the triple marker CKD tests not yet done(creatinine, urine microalbumin, cystatin C). Once the tests are ordered, patients will proceed to the laboratory as they normally would in clinical practice. The EHR will be programmed to return the results to the PCP's clinical results folder in APeX, and to a study inbox monitored by the study MDs. Participating PCPs will be advised about tests being ordered along with a list of their eligible patients when sent the opt out letter prior to being randomized.

Best Practice Alert (BPA), Smart Set: The CDSS will allow a "second-chance" for test ordering if the tests are not completed prior to an enrolled patient encounter (for PCPs in the CDSS or CDSS Plus arms), by automatically delivering a reminder message embedded in the visit encounter as part of a best practice alert (BPA) indicating that the triple marker tests have been ordered but not completed for this patient. If the tests have been completed at the time of the visit, the BPA will give CKD staging based on the triple marker for the individual patient and have a button to click to open a smart smart-set tailored to that specific patient. The smart-set will cover the orders and recommendations as indicated for that patient: Blood pressure target, use of ACEI/ARB class of medications, potassium management, use of statin medications, pre-populated referral to nephrology when indicated, patient educational material on NSAIDS and CKD in general to populate the After Visit Summary.

CDSS PLUS: The rationale for this third arm is based on the evidence that clinical pharmacists have been shown to be more effective than physicians alone at achieving BP control in other settings. For PCPs in the CDSS PLUS intervention arm, the study will provide cards identifying the pharmacist on the clinical team. During the visit in which the CDSS launches, the PCPs can let the patient know that a pharmacist, who is part of the clinical team, will be calling to follow-up, and he/she can hand these cards out to eligible patients. In addition, the CDSS smart set for these patients will give information about the pharmacist that can populate the After Visit Summary. This warm hand-off will allow the patient to be aware of the reason for the pharmacist's post-visit call. For patients active on MyChart, the pharmacist will use MyChart to set up a good time to call the patient within two weeks. If the patient does not use MyChart, the pharmacist will attempt to call and leave messages for the patient. On the phone call, the pharmacist will discuss and collect data on the patient's understanding of CKD, conduct a medication review and adherence assessment, ask about home BP checks, and discuss the importance of NSAID avoidance.

All calls will be documented in APeX to allow the entire clinical team to follow the patient's care and route messages to the PCP and team RN as necessary. A second call from the pharmacist will only be triggered if the patient is non-adherent and makes an active plan for adherence requiring a follow-up call to check-in on that plan, or if the patient requests an additional follow-up call.

ELIGIBILITY:
Inclusion Criteria:

* Have at least two outpatient, documented eGFRcreat values 30- 59 ml/min/1.72m2 that are at least ≥3 months apart
* At least one of these measurements should be within 12 months.
* Patients have seen their primary care physician at least one time within the previous 18 months
* Patient's primary care providers agree to participate

Exclusion Criteria:

* Patients actively and recently seen by nephrology clinic (at least once in the past 12 months)
* Patients with a diagnosis of end stage renal disease
* Persons aged >80
* Persons with New York Heart Association (NYHA) class III or IV heart failure, known ejection fraction < 25%, or documented allergy to ace/arb.
* Patients on dialysis, kidney transplant recipients and pregnant women
* Patients with prevalent dementia, impaired cognition or severe mental illness; expected life expectancy < 6 months.

There will also be a category where the physician can opt out for specific patients in their panel due to not believing this person should be included in the study for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from enrollment | Investigators will follow patients up to 2 years after measures
  Clinical Outcome: The primary clinical outcome of the trial is change in blood pressure (mmHg) from enrollment to the end of the follow up period as a continuous outcome, ascertained from the electronic medical record. BP measures from the clinical record will be ascertained in no more than quarterly intervals in the primary care setting to avoid bias by ascertainment. Investigators will also consider the dichotomous clinical outcome "achieved sustained BP control", defined as BP < 140/90 mmHg in ≥ two consecutive visits during the trial.

SECONDARY OUTCOMES:
Feasibility | Investigators will follow patients up to 2 years after measures
  Investigators will assess provider awareness of CKD, defined as percent appropriate inclusion of CKD in the problem list (dichotomous outcome).
Processes of Care | Investigators will follow patients up to 2 years after measures
  Investigators will also measure use of ACEI/ARB among persons with albuminuria, measured as the proportion (percent) of persons on these medications at the end of the study period, compared to enrollment. Medication prescription will be ascertained by percent with an electronic record of a new order or modification during the study period, not including refills. Other process outcomes relate to feasibility and the ability to implement the CDSS protocol. These include proportion in the intervention arms with completion of albuminuria and cystatin C testing.
CKD and NSAID avoidance Knowledge | Investigators will interview each participant 2 weeks after their primary care visit or clinical pharmacist phone call
  Patient-centered outcomes: Investigators will evaluate CKD and NSAID avoidance knowledge (proportion with correct answers), using structured telephone interviews, and comparing patients from the three study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Division of General Internal Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Plan for monitoring data and safety: A recommendation to order a creatinine and potassium level following initiation or up-titration of ace/arb will be incorporated in the algorithm in the result note. A 24/7 line to a nephrology answering service will be available to participating Primary Care Providers (PCPs) in the case of critical results; for non-critical study-related questions, participating PCPs can contact the study nephrologist via staff messaging in APeX. If a patient is found to have eGFR < 30 ml/min/1.73m2, investigators will recommend nephrology referral for pre-dialysis care.

REFERENCES:
- [Result] Coresh J, Byrd-Holt D, Astor BC, Briggs JP, Eggers PW, Lacher DA, Hostetter TH. Chronic kidney disease awareness, prevalence, and trends among U.S. adults, 1999 to 2000. J Am Soc Nephrol. 2005 Jan;16(1):180-8. doi: 10.1681/ASN.2004070539. Epub 2004 Nov 24. PMID 15563563
- [Result] Peralta CA, Shlipak MG, Judd S, Cushman M, McClellan W, Zakai NA, Safford MM, Zhang X, Muntner P, Warnock D. Detection of chronic kidney disease with creatinine, cystatin C, and urine albumin-to-creatinine ratio and association with progression to end-stage renal disease and mortality. JAMA. 2011 Apr 20;305(15):1545-52. doi: 10.1001/jama.2011.468. Epub 2011 Apr 11. PMID 21482744
- [Result] Shlipak MG, Coresh J, Gansevoort RT. Cystatin C versus creatinine for kidney function-based risk. N Engl J Med. 2013 Dec 19;369(25):2459. doi: 10.1056/NEJMc1312801. No abstract available. PMID 24350959
- [Result] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Derived] Peralta CA, Livaudais-Toman J, Stebbins M, Lo L, Robinson A, Pathak S, Scherzer R, Karliner LS. Electronic Decision Support for Management of CKD in Primary Care: A Pragmatic Randomized Trial. Am J Kidney Dis. 2020 Nov;76(5):636-644. doi: 10.1053/j.ajkd.2020.05.013. Epub 2020 Jul 22. PMID 32682696
- [Derived] Khoong EC, Karliner L, Lo L, Stebbins M, Robinson A, Pathak S, Santoyo-Olsson J, Scherzer R, Peralta CA. A Pragmatic Cluster Randomized Trial of an Electronic Clinical Decision Support System to Improve Chronic Kidney Disease Management in Primary Care: Design, Rationale, and Implementation Experience. JMIR Res Protoc. 2019 Jun 7;8(6):e14022. doi: 10.2196/14022. PMID 31199334